CLINICAL TRIAL: NCT05251129
Title: Statin InTensity to Prevent Coronary Artery Vasculopathy After Heart Transplantation - SToP-CAV
Brief Title: Statin InTensity to Prevent Coronary Artery Vasculopathy After Heart Transplantation
Acronym: SToP-CAV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never submitted. Study team instead conducted a retrospective study which did not qualify for registration.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-13700
Record Dates: First submitted 2021-12-17; First posted 2022-02-22 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Vasculopathy
MeSH Terms: conditions — Vascular Diseases | interventions — Atorvastatin; Tablets; Pravastatin

STUDY DESIGN:
Intervention Model Description: Open-label, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher Intensity Statin (Experimental): Atorvastatin 80 milligram (mg) oral tablet
  Interventions: Drug: Atorvastatin 80 Mg Oral Tablet
- Lower Intensity Statin (Active Comparator): Pravastatin 40 mg oral tablet
  Interventions: Drug: Pravastatin 40 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 80 Mg Oral Tablet — Higher intensity statin
  Arms: Higher Intensity Statin
Drug: Pravastatin 40 Mg Oral Tablet — Lower intensity statin
  Arms: Lower Intensity Statin

SUMMARY:
The investigator's propose to conduct an open-label randomized controlled trial to determine if higher intensity statin (HS) can reduce CAV in comparison to lower intensity statin (LS) after HT. All consecutive patients that meet eligibility criteria will be approached for participation. After heart transplantation, participants (n=70) will be randomized in a 1:1 manner to either HS or LS. Study participation will be for 2 years from the time of randomization. Study outcomes will be compared by research staff blinded to statin group assignment.

DETAILED DESCRIPTION:
Outcomes after heart transplantation (HT) are limited by development of coronary allograft vasculopathy (CAV). CAV comprises of macro- and microvascular coronary disease and is the third leading cause of graft dysfunction and late mortality following HT. The pathophysiology of CAV is multifactorial and major pathways that are implicated include inflammation and dyslipidemia. These pathways are inhibited by statins which serve as the mainstay of CAV prevention.

The International Society of Heart and Lung Transplantation (ISHLT) guidelines recommend administration of low intensity statins (LS) due to a potential drug-drug interaction (DDI) with calcineurin inhibition (CNI) therapy. This DDI is related to concurrent use of an older generation CNI, cyclosporin A (CsA). CsA inhibits intestinal P-glycoprotein to reduce the efflux of statin into the gastrointestinal tract, thereby increasing statin levels in the blood and risk of myopathy. However, the current generation of CNI being utilized in most patients, Tacrolimus, does not inhibit P glycoprotein and may not impact statin levels after HT.

Despite use of LS, the residual risk of CAV development is elevated with nearly half of the patients having angiographic detection 5 years after HT. However, angiography is limited by its inability to detect microvascular disease and invasiveness. Early CAV is also detectable by non-invasive imaging with cardiac positron emission tomography (cPET) through measurement of myocardial flow reserve (MFR). MFR assesses total burden of macro- and microvascular disease and is well correlated with invasive measures of CAV and prognosis.

The protective and inhibitory effects of statins are proportional to their intensity with higher intensity statins (HS) leading to a greater reduction in low density lipoprotein (LDL) and inflammatory markers such as C-reactive protein (CRP) in comparison to LS. Despite these potentially beneficial effects of HS, LS remains the agent of choice for primary prevention of CAV after HT in the absence of a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Waitlisted for Heart Transplantation
* Capacity to provide informed consent

Exclusion Criteria:

* History of statin allergy or intolerance
* Hepatic dysfunction
* Redo Heart Transplant
* Awaiting combined heart and liver transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Myocardial Flow Reserve | 2 year
  Myocardial Flow Reserve measured by cardiac positron emission tomography

SECONDARY OUTCOMES:
Coronary Vascular Resistance | 2 year
  Coronary Vascular Resistance measured by cardiac positron emission tomography
Change in Global Longitudinal Strain | baseline, 1 year and 2 year
  Change in Global Longitudinal Strain measured by echocardiography
Blood level of Low Density Lipoprotein | baseline, 6, 12, 18, 24 months
  Blood level of Low Density Lipoprotein
Blood level of High Sensitivity C-Reactive Protein | baseline, 6, 12, 18, 24 months
  Blood level of High Sensitivity C-Reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: Omar Saeed, MD, MS, Principal Investigator — Montefiore Medical Center